CLINICAL TRIAL: NCT02933827
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of Allogeneic Infusion of Adipose-Derived Stem Cells in Moderate to Severe Chronic Kidney Disease
Brief Title: Adipose-derived Stem Cells (ADSCs) for Moderate to Severe Chronic Kidney Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UnicoCell Biomed CO. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT31
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2020-11

CONDITIONS: Moderate to Severe Chronic Kidney Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose: (Experimental): ELIXCYTE 8 mL (ADSC 6.4*10^7 cells in total)
  Interventions: Drug: ELIXCYTE
- Middle dose (Experimental): ELIXCYTE 24 mL (ADSC 19.2*10^7 cells in total)
  Interventions: Drug: ELIXCYTE
- High dose (Experimental): ELIXCYTE 40 mL (ADSC 32.0*10^7 cells in total)
  Interventions: Drug: ELIXCYTE

INTERVENTIONS:
Drug: ELIXCYTE — Adipose-derived stem cells (ADSCs)

SUMMARY:
1. To assess the safety of allogeneic injection of expanded ADSCs to patients with Moderate to Severe Chronic Kidney Disease
2. To assess the efficacy of allogeneic injection of expanded ADSCs to patients with Moderate to Severe Chronic Kidney Disease

ELIGIBILITY:
Inclusion Criteria:

A patient is eligible for the study if all of the followings apply:

1. Aged 20-80 years (inclusive)
2. With chronic kidney disease (CKD)stage 3B to 4 (eGFR 15 to 44 mL/min/1.73m2 (inclusive)) Note : eGFR = estimated glomerular filtration rate
3. Having provided informed consent

Exclusion Criteria:

Any patient meeting any of the exclusion criteria will be excluded from study participation.

1. Ascertained hypersensitivity to any component used in the study Note: including gentamicin, DMSO, Agglutex (heperin)
2. With inadequate hematologic function with: absolute neutrophil count (ANC) <1,500/μL OR platelets < 100,000/μL OR Hemoglobin < 8 g/dL
3. With inadequate hepatic function with: serum bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase (AKP) > 2.5 x the institutional upper limit of normal (ULN)
4. With hemoglobin A1c (HbA1c) > 8.0%
5. With serious prior or ongoing medical conditions (e.g. concomitant illness such as cardiovascular (e.g. New York Heart Association grade III or IV), hepatic (e.g. Child-Pugh Class C), psychiatric condition, alcoholism, drug abuse), medical history, physical findings, ECG findings, or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely affect the safety of the patient
6. Pregnant or lactating women or premenopausal with childbearing potential but not taking reliable contraceptive method(s) during the study period
7. With body mass index (BMI) greater or equal to 36 kg/m2
8. With known history of human immunodeficiency virus (HIV) infection or any type of hepatitis
9. Judged to be not applicable to this study by investigator such as difficulty of follow-up observation
10. With any other serious diseases/medical history considered by the investigator not in the condition to enter the trial
11. Having participated other investigational study within 4 weeks of entering this study
12. Known or suspected abuse of alcohol or narcotics
13. With known history of cancer within past 5 years
14. With any autoimmune disease
15. With cystic kidney disease or requiring kidney dialysis
16. With precancerous condition or with cancer within past 5 years before Screening visit

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Week 48
  for Phase I
Change from baseline to Week 24 visit in estimated glomerular filtration rate (eGFR) | Week 0, 24
  or Phase II

SECONDARY OUTCOMES:
Change from baseline to all post-treatment visits in creatinine | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in blood urea nitrogen (BUN) | Weeks 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in blood cystatin C | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in urine total protein-creatinine ratio (UPCR) | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in plasma neutrophil gelatinase-associated lipocalin (NGAL) by enzyme-linked immunosorbent assay (ELISA) | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in urine kidney injury molecule-1(KIM-1) | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in urine interleukin 18 (IL-18) | Weeks 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in urine liver-type fatty acid-binding protein (L-FABP) | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in urine neutrophil gelatinase-associated lipocalin (NGAL) | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in urine cystatin C | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in hemoglobin A1c | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in fasting plasma glucose | Weeks 0, 2, 4, 12, 24, 36, 48
Percentage of patients with hypoglycemia (defined as blood glucose < 55 mg/dL or 3.0 mmol/L) at all post-treatment visits | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in body weight | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in urine microalbumin-to-creatinine ratio (UMCR) | Weeks 0, 2, 4, 12, 24, 36, 48
Change from baseline to all post-treatment visits in eGFR | Weeks 0, 2, 4, 12, 24, 36, 48

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Szu Wu, PhD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (3):
- Taiwan (3):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Chang Gung Memorial Hospital Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin YC, Hung YP, Tian YC, Wu MJ, Lin HC, Chen SY, Wu MS, Chiou HY. Real-World Data as External Control in Assessing the Efficacy of Allogeneic Adipose-Derived Stem Cells Therapy for Advanced Chronic Kidney Disease. Clin Transl Sci. 2025 Dec;18(12):e70415. doi: 10.1111/cts.70415. PMID 41299839
- [Derived] Zheng CM, Chiu IJ, Chen YW, Hsu YH, Hung LY, Wu MY, Lin YF, Liao CT, Hung YP, Tsai CC, Cherng YG, Wu MS. Allogeneic adipose tissue-derived stem cells ELIXCYTE(R) in chronic kidney disease: A phase I study assessing safety and clinical feasibility. J Cell Mol Med. 2022 May;26(10):2972-2980. doi: 10.1111/jcmm.17310. Epub 2022 Apr 12. PMID 35415928